CLINICAL TRIAL: NCT01462149
Title: Phase II Trial of Docetaxel and Carboplatin as Neoadjuvant Chemotherapy in Patients With Advanced Ovarian Cancer
Brief Title: Efficacy Study of Neoadjuvant Chemotherapy to Treat Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Jong-Hyeok Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEODOCA-OVCA
Record Dates: First submitted 2011-10-25; First posted 2011-10-31 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Advanced Ovarian Cancer
MeSH Terms: interventions — Neoadjuvant Therapy; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy (Experimental): Neoadjuvant chemotherapy with docetaxel plus carboplatin
  Interventions: Drug: Neoadjuvant chemotherapy; Drug: Carboplatin

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy — Docetaxel 75mg/m2BAS, q 3 weeks, 3 cycles
Drug: Carboplatin — Carboplatin AUC 5, q 3 weeks, 3 cycles

SUMMARY:
Neoadjuvant chemotherapy is alternative treatment option to upfront cytoreductive surgery to treat advanced ovarian cancer. Paclitaxel plus carboplatin is most frequently selected chemotherapeutic regimen for neoadjuvant chemotherapy. Docetaxel had similar therapeutic efficacy compared to paclitaxel in adjuvant chemotherapy trials in ovarian cancer. However, docetaxel had more favorable toxicity profile. Therefore, the investigators aimed to evaluate the efficacy of docetaxel plus carboplatin as neoadjuvant chemotherapy in patients with advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced epithelial, tubal, or primary peritoneal cancer
* Cancer cells in paracentesis, thoracentesis, or laparoscopic surgery
* Less probability of complete cytoreduction
* Age: 20-80 years
* GOG performance status: 0-3
* Adequate organ function Bone marrow: ANC ≥ 1,500mm3, Platelet ≥ 100,000/mm3, Hb ≥ 10.0 g/dl Kidney: Creatinine ≤ 1.25 × UNL Liver: AST, ALT ≤ × 2.5 UNL (in case of liver metastasis, AST, ALT ≤ × 5 UNL), alkaline phosphatase ≤ 5 x UNL, bilirubin ≤ 1.5 mg/ mm3

Exclusion Criteria:

* Previous chemotherapy or pelvic radiation therapy
* Final diagnosis is other malignancies
* Coincidental Other malignancies within 5 years except carcinoma in situ of uterine cervix
* History of severe allergy
* Pregnancy, lactating woman
* Uncontrolled medial disease
* Bowel obstruction requiring immediate surgery
* Etc.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Response rate | 1 month after completion of study treatment

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Before each chemotherapy, an average of 3 week
Disease-free survival | 2 years after completion of study treatment
Overall survival | 2 years after completion of study treatment
The number of participants who achieved optimal cytoreduction | 1 month after completion of study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea